

#### Informed Consent and HIPAA Authorization Form

Study Title: Investigating the experience of living with Down Syndrome and

obstructive sleep apnea syndrome

Version Date: August 2, 2019

**Principal Investigator:** Ignacio Tapia, MD Telephone: (215) 590-3749

You and your child may be eligible to take part in a research study. This form gives you important information about the study. It describes the purpose of this research study, and the risks and possible benefits of participating.

In the sections that follow, the word "we" means the study doctor and other research staff. If you are a parent or legal guardian who is giving permission for a child, please note that the word "you" refers to your child.

# **Study Overview**

You and your parent are being asked to take part in this research study because your child has Down syndrome and obstructive sleep apnea.

The purpose of this research study to learn more about the experience of living with Down syndrome and obstructive sleep apnea.

If you take part, you will be asked to:

- Have your medical records reviewed
- Your parent will participate in a 30 minute phone audio-recorded interview

The main risks of this study are from the recorded interview. These include a breach of confidentiality.

You will not benefit directly from participating in this study

Participation in this study is voluntary. If you do not choose to take part in this study, you can discuss other options with your doctor.

If there is anything in this form you do not understand, please ask questions. Please take your time. You do not have to take part in this study if you do not want to. If you take part, you can leave the study at any time.

If you are interested in learning more about the study, please continue to listen.

CHOP IRB#: IRB 19-016222 Effective Date: 8/2/2019

Expiration Date: N/A

Page 1 of 6

# What are the study procedures?

Medical Record Review: We will review your medical records to collect information about your medical history, sleep study results, and information related to your PAP use and diagnoses

<u>Interview</u>: We will ask your parent to complete one semi-structured interview over the phone. The interview will be audio-recorded.

# What are the risks of this study?

Taking part in a research study involves inconveniences and risks. The main risks of taking part in this study are discussed below.

#### **Risk of Recorded Interviews**

The main risk to you is that someone could find out you were in this study. But we will do our best to keep your information confidential, so we think this risk is very low. Some people may feel uncomfortable having the interview recorded. You may skip any question or stop the interview at any time.

# Risk of Breach of Confidentiality

As with any study involving collection of data, there is the possibility of breach of confidentiality of data. Every precaution will be taken to secure participants' personal information to ensure confidentiality. At the time of participation, each participant will be assigned a study identification number. This number will be used on data collection forms and in the database instead of names and other private information. A separate list will be maintained that will links each participant's name to the study identification number for future reference and communication.

# Are there any benefits to taking part in this study?

There will be no direct benefit to you from taking part in this study. The knowledge gained from this study may help doctors know more about the experience of living with DS and OSAS.

# Do you need to give your consent in order to participate?

If you decide to participate in this study, you must tell us that you agree. A copy will be given to you to keep as a record.

#### What are your responsibilities?

Please consider the study time commitments and responsibilities as a research subject when making your decision about participating in this study.

#### What happens if you decide not to take part in this study?

Participation in this study is voluntary. You do not have to take part in order to receive care at CHOP.

If you decide not to take part or if you change your mind later there will be no penalties or loss of any benefits to which you are otherwise entitled.

CHOP IRB#: IRB 19-016222 Effective Date: 8/2/2019

Expiration Date: N/A

#### Can you stop your participation in the study early?

You can stop being in the study at any time. You do not have to give a reason.

### Can the study doctor take you out of the study early?

The study doctor may take you off of the study if:

- You repeatedly fail to keep your phone interview appointment
- The study is stopped.

# What about privacy, authorization for use of Personal Health Information (PHI) and confidentiality?

As part of this research, health information about you will be collected. This will include information from medical records, and interviews. Information that could identify you will not be shared with anyone - unless you provide your written consent, or it is required or allowed by law. We will do our best to keep your personal information private and confidential. However, we cannot guarantee absolute confidentiality. Your personal information may be disclosed if required by law.

The results of this study may be shown at meetings and published in journals to inform other doctors and health professionals. We will keep your identity private in any publication or presentation.

Several people and organizations may review or receive your identifiable information. They will need this information to conduct the research, to assure the quality of the data, or to analyze the data or samples. These groups include:

- Members of the research team and other authorized staff at CHOP
- Mixed Methods Research Lab at the University of Pennslyvania
- The National Institutes of Health who is sponsoring this research;
- People from agencies and organizations that perform independent accreditation and/or oversight of research; such as the Department of Health and Human Services, Office for Human Research Protections.

By law, CHOP is required to protect your health information. The research staff will only allow access to your health information to the groups listed above. By telling us that you agree, you are authorizing CHOP to use and/or release your health information for this research. Some of the organizations listed above may not be required to protect your information under Federal privacy laws. If permitted by law, they may be allowed to share it with others without your permission.

The identifiable information from this study will be destroyed 6 years after the study is completed. Your permission to use and share the information and data from this study will continue until the research study ends and will not expire. Researchers continue to analyze data for many years and it is not possible to know when they will be completely done.

# **Certificate of Confidentiality (CoC)**

CHOP IRB#: IRB 19-016222 Effective Date: 8/2/2019 Expiration Date: N/A **3**H

A Certificate of Confidentiality (CoC) covers this research. A CoC helps protect your identifiable information.

A CoC protects your private information from all legal proceedings. Unless you consent, information from this research study that identifies you will not be shared outside this research.

- No one can be forced to share your identifiable information or biological samples for a lawsuit.
- Your information can't be used as evidence even if there is a court subpoena.

If you consent, your data could be shared for:

• other scientific research;

The CoC does not prevent some disclosures.

- The researchers can't refuse requests for information from those funding this
  research. The National Institutes of Health may need information to assess this
  project.
- You can still share information about yourself. You can also freely discuss your involvement in this research.
- The researchers must disclose things required by law. This includes suspected child abuse and neglect, harm to self or others, or communicable diseases.

# Can you change your mind about the use of personal information?

You may change your mind and withdraw your permission to use and disclose your health information at any time. To take back your permission, it is preferred that you inform the investigator in writing.

Dr. Ignacio Tapia Children's Hospital of Philadelphia Division of Pulmonary Medicine 34<sup>th</sup> Street and Civic Center Blvd. Philadelphia, PA 19104

In the letter, state that you changed your mind and do not want any more of your health information collected. The personal information that has been collected already will be used if necessary for the research. No new information will be collected. If you withdraw your permission to use your personal health information, you will be withdrawn from the study.

#### **Financial Information**

Will there be any additional costs?

There will be no additional costs to you by taking part in this study.

Will you be paid for taking part in this study?

CHOP IRB#: IRB 19-016222 Effective Date: 8/2/2019

Effective Date: 8/2/2019 Expiration Date: N/A



• Participants will be paid \$50.00 gift card for their time and effort after the phone interview is completed.

# Who is funding this research study?

The National Institutes of Health is funding this research.

# What if you have questions about the study?

If you have questions about this study or how your data are going to be used, call the study doctor, Dr. Tapia at 215-590-3749. You may also talk to your own doctor if you have questions or concerns.

The Institutional Review Board (IRB) at The Children's Hospital of Philadelphia has reviewed and approved this study. The IRB looks at research studies like these and makes sure research subjects' rights and welfare are protected. If you have questions about your rights or if you have a complaint, you can call the IRB Office at 215-590-2830.

# What will be done with my data when this study is over?

We will use and may share data for future research. They may be shared with researchers/institutions outside of CHOP. This could include for profit companies. We will not ask for your consent before using or sharing them. We will remove identifiers from your data, which means that nobody who works with them for future research will know who you are. Therefore, you will not receive any results or financial benefit from future research done on your data.



CHOP IRB#: IRB 19-016222 Effective Date: 8/2/2019 Expiration Date: N/A

# Documentation of Verbal Consent to Take Part in this Research Study and Authorization to Use and Disclose Health Information for the Research

| Name of Child Subject | Name of Parent Subject |
|---|---|
| The research study and consent form | was explained to: |
| Person Providing Consent | Relation to child subject: Parent Legal Guardian |
| 1 1 | nfirmed that all of their questions had been ir child's participation in this research study. |
| They confirmed that they were legally participation. | y authorized to consent to their child's |
| They agreed to let CHOP use and sha | re their child's health information. |
| Person Obtaining Consent | Signature of Person Obtaining Consent |
| | Date |



Expiration Date: N/A

